CLINICAL TRIAL: NCT06672796
Title: Comparison of the Effects of Standard and Resisted Protocols of Toe Spread Out Exercise on Hallux Valgus Angle, Muscular Activation, Balance and Physical Performance in Individuals with Hallux Valgus.
Brief Title: Comparison of the Effects of Different Exercise Protocols in Individuals with Hallux Valgus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahar Anaforoglu (Other)
Responsible Party: Sponsor-Investigator, Bahar Anaforoglu, Associate Professor, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AnkaraYbu2024HV
Record Dates: First submitted 2024-10-30; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Hallux Valgus Deformity
Keywords: hallux valgus; toe spread out; physiotherapy; ultrasound; surface electromyography
MeSH Terms: conditions — Hallux Valgus | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Randomised controlled
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CG (Active Comparator): 8 weeks, stretching exercise
  Interventions: Other: Stretching exercise
- SEG (Active Comparator): 8 weeks, stretching exercise and toe spread out standart protocol
  Interventions: Other: Toe Spread Out Exercise; Other: Stretching exercise
- REG (Experimental): 8 weeks, stretching exercise and resisted concentric and eccentric contraction protocol of toe spread out exercise
  Interventions: Other: Resisted Toe Spread Out Exercise; Other: Stretching exercise

INTERVENTIONS:
Other: Resisted Toe Spread Out Exercise — new resistance exercise phase in addition to the standard protocol
  Arms: REG
Other: Toe Spread Out Exercise — Standart protocol of toe spread out exercise
  Arms: SEG
Other: Stretching exercise — Toe stretching

SUMMARY:
The aim of this study was to determine the effects of 8 weeks of supervised in addition to stretching exercise resisted concentric and eccentric contraction protocol of toe spread out exercise on the angular severity of hallux valgus deformity, changes in the cross-sectional area, stiffness and thickness of the abductor hallucis muscle, electromyographic activities, plantar pressure distribution, foot morphology and gait characteristics, balance and physical performance at the end of the medium and long term.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65,
* Being diagnosed with mild or moderate HV according to the radiographic evaluation result,
* Having flexible HV,
* Being a volunteer

Exclusion Criteria:

* Having a neurological disease,
* Having a systemic disease,
* Having cognitive disorders such as dementia, Alzheimer's, etc.,
* Having spinal problems such as disc herniation, lumbar stenosis, scoliosis, etc.,
* Having claudication,
* Having idiopathic numbness, tingling, etc. complaints in the lower extremity,
* Having had lower extremity surgery before,
* Having a fracture, ligament, or muscle injury in the lower extremity within the last 6 months,
* Having received foot-related treatment within the last 6 months.
* Not understanding the exercises,
* Not being able to continue with exercise sessions,
* Low homework exercise compliance,
* Foot structure not suitable for elastographic US examination,
* Incorrectly measured elasticity values in SWE,
* Not participating in the first or last evaluation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Hallux Valgus Angle | Before treatment, after 6 months
  A radiographic measurement (°) The angle created between the lines that longitudinally bisect the proximal phalanx and the first metatarsal.
Intermetatarsal angle | Before treatment, after 6 months
  A radiographic measurement (°) The term intermetatarsal angle alone typically refers to assessment of the first and second metatarsals
Hallux Interphalangeal Angle | Before treatment, after 6 months
  A radiographic measurement (°) The hallux interphalangeal angle is between the proximal and distal phalanx of the great toe and serves for the evaluation of toe deformity at the level of the first interphalangeal joint.
Distal Metatarsal Articular Angle | Before treatment, after 6 months
  A radiographic measurement (°) The distal metatarsal articular angle (DMAA) evaluates the relationship between the longitudinal axis and the articular surface of the first metatarsophalangeal joint and thus metatarsophalangeal coverage or joint congruity on a weight-bearing dorsoplantar radiograph of the foot.
Sesamoid Position Classification | Before treatment, after 6 months
  A radiographic measurement (1-7 grades) The medial sesamoid position would be classified into 7 grades by the respective circle as the position of the medial sesamoid.
Length of the First Metatarsal | Before treatment, after 6 months
  A radiographic measurement Length of the first metarsal (centimeter)
Surface Electromyography | Before first treatment, after 8 weeks, and after 6 months
  Maximum volunteer isometric contarction (MVIC) of m. abductor hallucis
Cross Sectional Area | Before treatment, after 8 weeks, after 6 months
  CSA of m. abductor hallucis with ultrasound (cm²) CSA: In muscle physiology, physiological cross-sectional area (PCSA) is the area of the cross section of a muscle perpendicular to its fibers, generally at its largest point
Dorsoplantar Thickness | Before treatment, after 8 weeks, after 6 months
  Measurement muscle thickness (m. abductor hallucis) with ultrasound (cm)
Mediolateral Width | Before treatment, after 8 weeks, after 6 months
  Measurement muslce width (m. abductor hallucis) with ultrasound (cm)
Shear Wave Elastography | Before treatment, after 8 weeks, after 6 months
  Measurement SWE with ultrasound (m. abductor hallucis) (cm)
Plantar load | Before treatment, after 8 weeks, after 6 months
  Measurement with plantar pressure distrubiton analysis (kg/cm²)
Loads per unit of plantar segments | Before treatment, after 8 weeks, after 6 months
  Measurement with plantar pressure distrubiton analysis (kg/cm²)
Changes of loads during gait | Before treatment, after 8 weeks, after 6 months
  Measurement with plantar pressure distrubiton analysis (kg/cm²)
Gait-time graph | Before treatment, after 8 weeks, after 6 months
  Measurement with plantar pressure distrubiton analysis (%)
Maximum and average pressures | Before treatment, after 8 weeks, after 6 months
  Measurement with plantar pressure distrubiton analysis (kg/cm²)
Plantar Contact area | Before treatment, after 8 weeks, after 6 months
  Measurement with plantar pressure distrubiton analysis (cm²)
Plantar contact time | Before treatment, after 8 weeks, after 6 months
  Measurement with plantar pressure distrubiton analysis (msn)
Balance measurement | Before first treatment, after 8 weeks, and after 6 months
  Y-balance test
Physical performance tests | Before first treatment, after 8 weeks, and after 6 months
  Gait speed (10 meter), Climbing stairs speed (10 meter)
Multidimensional Nil Hallux Valgus Scale | Before first treatment, after 8 weeks, and after 6 months
  The scale has a score range of 0-60, with higher score indicating increased HV symptoms, complaints, and functional disorder.